CLINICAL TRIAL: NCT05834959
Title: Implementation of a Fitness Education and Training Program to Support Safe Patient Handling and Safe Lifting in a Community Based Hospital (The Fit for Work Project)
Brief Title: Implementation of a Fitness Education and Training Program to Support Safe Patient Handling and Safe Lifting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: The Wellness Institute Powered by Seven Oaks General Hospital (Unknown); Workers Compensation Board of Manitoba (Unknown); Seven Oaks General Hospital (Unknown)
Responsible Party: Principal Investigator, Shelley Sargent, Manager of Patient Care-Rehab Physiotherapy, PAR Health Services and Child Health, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS25745 (H2022:355)
Record Dates: First submitted 2023-03-13; First posted 2023-04-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lower Back Injury
Keywords: Safe Patient Handling; Safe Lifting; Injury Prevention.; Program Outcome Evaluation

STUDY DESIGN:
Intervention Model Description: A two-part education and practical program designed to evaluate the effects of training on movement confidence, low back dysfunction and changes in rates of lower back injury. SPSS software will be used to analyze mean differences between self-report questionnaire scores regarding low back pain/dysfunction at baseline and post-program using paired t-tests (p<0.05). Paired t-tests will be used to determine if there is a statistical difference in back injury rates at Seven Oaks Hospital one year post-program, compared to previous years. The results of the post-program survey will be summarized using descriptive statistics. Information from baseline movement confidence questionnaires will also be summarized using descriptive statistics and compared pre and post programming.
  *Note: Before t-test analyses is performed the distribution of scores will be checked to determine if they are normal. If not, non-parametric tests equivalent to paired t-tests will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOGH employees, taking part in the same education and training program. (Experimental): Participants will be recruited from the Seven Oak General Hospital staff population and will complete a two-part education and practical program.
  Interventions: Other: An Educational and Training Program

INTERVENTIONS:
Other: An Educational and Training Program — Education and practical training program designed to evaluate the effects of training on movement confidence, low back dysfunction and changes in rates of lower back injury

SUMMARY:
This project involves the delivery of education and training sessions to Seven Oaks General Hospital (SOGH) staff, with the goal of workplace injury prevention. Education will include review of provincial safe patient handling and back injury prevention guidelines and review of core fitness competencies required to comply with injury prevention standards. Training sessions will include exercises to improve core, gluteal and quadricep strength, hip/knee mobility and hamstring flexibility. Training will also be an opportunity to provide feedback on functional movement performance. Outcomes will include questionnaires on: low back pain/dysfunction; movement confidence; work injury rates and participant satisfaction with program. The project will advise stakeholders of the benefits and challenges associated with implementation of a fitness program to support safe patient handling techniques, as outlined in the provincial guidelines for healthcare workers.

DETAILED DESCRIPTION:
The Fit for Work Project is an educational and training program outcome evaluation. It is a two-part education and practical program designed to evaluate the effects of training on movement confidence, low back dysfunction and changes in rates of lower back injury. In the first part, participants will attend the education session developed by physiotherapists who specialize in return to work programs. In the second part participants will participate in a 4-week practical program, where they will stretch, lengthen and strengthen key muscles used in squatting, weight shifting and the hip hinge movement. Feedback and movement coaching are an important element in performing and mastering these movements correctly and this workplace wellness training program will provide staff the support needed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older
* Staff of Seven Oaks General Hospital during the time of the program
* Able to communicate in English and provide written informed consent

Exclusion Criteria:

* An acute injury, a medical condition, or other personal reason inhibiting participation in all 4 weeks of exercise training sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in staff confidence in performing the core fitness competencies required to abide by safe patient handling, safe lifting and back injury prevention guidelines | At the beginning of the program (baseline), at week 4 (the end of the 4-week training program), and one year after completion of the training program
  A Movement Confidence Questionnaire will be used, asking participants to rate their confidence as either 1-Very Low, 2-Low, 3-Moderate, 4-High, 5-Very High in completing 10 different movements without difficulty:
  1. Get down to and back up from the floor without using support
  2. Walk continuously for 1 hour
  3. Balance on 1 foot for 30 seconds
  4. Bend over to clean the bath tub
  5. Move the fridge to clean behind it
  6. Lift a 24 pack of water bottles off the floor
  7. Place carry-on luggage in overhead bin on airplane
  8. Lift a heavy suitcase in and out of the trunk of a car.
  9. Carry 2 heavy bags of groceries 100 ft or 30 m
  10. Shovel snow from a 1 car driveway.
Change from baseline in severity of low back pain and/or dysfunction | At the beginning of the program (baseline), at week 4 (the end of the 4-week training program), and one year after completion of the training program
  Measured as change from baseline in the Quebec Back Pain Disability Scale (Designed to evaluate functional limitations related to pain, to monitor the progress of individual patients and to compare the evolution of lower back pain (LBP) subjects incorporated in rehabilitation programs)
Change from baseline in severity of low back pain and/or dysfunction | At the beginning of the program (baseline), at week 4 (the end of the 4-week training program), and one year after completion of the training program
  Measured as change from baseline in the Oswestry Disability Index, also known as the Oswestry Low Back Pain Disability Questionnaire. (A self-reported measurement tool that measures both pain and functional status. It is used for evaluating disability caused by lower backache).
Change from baseline in incidence of back injuries | At the beginning of the program (baseline), and 1 year after completion of the 4-week training program
  Measured as change in the number of new low back injuries or flare-ups of existing back conditions sustained in the past year.
Change from baseline in frequency of back injuries | At the beginning of the program (baseline), and 1 year after completion of the 4-week training program
  Measured as the number of new low back injuries or flare-ups of existing back conditions sustained at work in the past year.
Change from baseline in time loss cost of back injuries | At the beginning of the program (baseline), and 1 year after completion of the 4-week training program
  Measured as the duration of time away from work due to low back pain/injury.

SECONDARY OUTCOMES:
Benefits and challenges associated with implementation of a fitness program to support safe patient handling and safe lifting techniques, as outlined in the provincial and regional guidelines for healthcare workers | Collected at week 4 (at the end of the 4-week training program)
  A "Program Exit Questionnaire" will be administered to collect participant experiences and views on the benefits and challenges associated with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Sargent, BMRPT MSc, Principal Investigator — The Wellness Institute at Seven Oaks General Hospital
Locations (1):
- The Wellness Institute, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No